CLINICAL TRIAL: NCT05806099
Title: A Phase I/Ⅱ Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Efficacy of MBS303 in Patients With Relapsed/Refractory B-Cell Non-Hodgkin's Lymphoma
Brief Title: A Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Efficacy Study of MBS303 in B-Cell NHL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing Mabworks Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MBS303-CT101
Record Dates: First submitted 2023-03-23; First posted 2023-04-10 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-07

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MBS303 (Experimental)
  Interventions: Drug: MBS303

INTERVENTIONS:
Drug: MBS303 — Phase I: The patients confirming to the eligibility criteria will be assigned to one of the 7 dose groups (0.05/0.15/0.45 mg ~ 1.5/6/60 mg, respectively) based on the sequence of inclusion. Each patient will receive MBS303 as per the schedule specified in the respective arms. Based on the safety data of the previous dose groups, if pretreatment with MIL62 is required after disussion by the sponsor and the investigators, the subject should be given an IV infusion of MIL62 1000 mg single dose on the D-7.
  Phase Ⅱ: One or two recommended doses will be selected based on the results of Phase I. Each patient will receive one of the two recommended doses MBS303 as step-up doses on D1 (low dose) and D8 (intermediate dose) of C1 and at the target dose on D1 of C2-17 (21-day cycles). Based on the previous safety data, if pretreatment with MIL62 is required after disussion by the sponsor and the investigators, the subjects should be given an IV infusion of MIL62 1000 mg single dose on the D-7

SUMMARY:
This is a Phase I/Ⅱ, multicenter, open-label, dose-escalation study designed to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics(PD) and efficacy of a novel T-Cell bispecific (TCB), MBS303, administered by intravenous (IV) infusion in participants with relapsed or refractory B-cell NHL. This entry-to-human study consists of 2 parts: a dose escalation part (Phase I) and an expansion part (Phase Ⅱ)

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent and to comply with the study protocol.
2. Adult patients, ≥18 years of age;
3. CD20+ B-cell Non-Hodgkin Lymphoma who have relapsed after or failed to respond to at least one prior treatment regimen with an anti-CD20 monoclonal antibody and for whom there is no available therapy expected to improve survival;
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
5. Life expectancy ≥3 months;
6. Measurable disease, defined as at lease one bi-dimensionally measurable nodal lesion, defined as >1.5 cm in its longest dimension, or at least one bi-dimensionally measureable extranodal lesion, defined as >1.0 cm in its longest dimension
7. Adequate hematologic, hepatic, and renal function.

Exclusion Criteria:

1. Chronic lymphoblastic leukemia, Burkitt lymphoma or lymphoplasmacytic lymphom;
2. History of central nervous system (CNS) lymphoma or other CNS disease;
3. Participants with known active infection, including bacterial, viral, parasite, mycobacterial, or other infections (excluding nail bed fungal infections);
4. Surgery, chemotherapy, targeted therapy, immunotherapy, radiation therapy, tumor embolization, or other antitumor therapy within 28 days prior to the first MBS303;
5. Active or suspected autoimmune diseases;
6. Known severe allergic reaction or/and infusion reaction to monoclonal antibody;
7. Evidence of significant, uncontrolled concomitant disease;
8. Major surgery within 28 days prior to the first MBS303 administration or expected to undergo major surgery during the study treatment;
9. History of another invasive malignant tumors in past 3 years;
10. Participant with history of confirmed progressive multifocal leukoencephalopathy (PML);
11. Severe hemorrhagic diseases such as hemophilia A, hemophilia B, vascular hemophilia, or spontaneous bleeding requiring blood transfusion or other medical intervention;
12. Infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C (including HBsAg, HBcAb positive with abnormal HBV DNA or HCV RNA);
13. Pregnant or lactating women; Females of childbearing potential (FCBP) must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual contact during the following time periods related to this study: 1) while participating in the study; 2) for at least 12 months after discontinuation of all study treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Phase I：Percentage of Participants with Adverse Events (AEs) | From Baseline up to approximately 13 months
  Percentage of Participants with AEs and SAEs Assessed by NCI CTCAE v5.0
Phase I：Incidence of Dose Limiting Toxicities (DLTs) | From Baseline up to 3 weeks
Phase I：Maximum Tolerated Dose (MTD) of MBS303 | From Baseline up to 3 weeks
Phase I：Recommended Phase Ⅱ Dose (RP2D) of MBS303 | From Baseline up to 4 years
Phase Ⅱ ：Antitumor activity as measured by the objective response rate (ORR) | Up to approximately 2 years

SECONDARY OUTCOMES:
Phase I and Ⅱ ：Pharmacokinetics: AUC | up to approximately 1 year
  The area under the curve (AUC) of serum concentration of MBS303 after the administration
Phase I and Ⅱ ：Pharmacokinetics: t1/2 | up to approximately 1 year
  Half-life (t1/2) of MBS303 after administration
Phase I and Ⅱ ：Pharmacokinetics: CL | up to approximately 1 year
  Clearance (CL) of MBS303 after administration
Phase I and Ⅱ ：Pharmacokinetics: Vd | up to approximately 1 year
  Volume of distribution (Vd) of MBS303 after administration
Phase I and Ⅱ ：Efficacy: Complete Response Rate (CRR) of MBS303 as Assessed Using Standard Criteria for NHL | Up to approximately 2 years
Phase I and Ⅱ ：Efficacy: Duration of Response (DOR) of MBS303 as Assessed Using Standard Criteria for NHL | Up to approximately 2 years
Phase I and Ⅱ ：Efficacy: Progression-Free Survival (PFS) of MBS303 as Assessed Using Standard Criteria for NHL | Up to approximately 2 years
Phase I and Ⅱ ：Efficacy: Overall Survival (OS) of MBS303 | Up to approximately 2 years
Phase I and Ⅱ ：Immunogenicity: Anti-Drug Antibodies (ADA) to MBS303 | Up to approximately 1 year
Phase I :Efficacy: ORR | Up to approximately 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China